CLINICAL TRIAL: NCT00585585
Title: A Pilot Study of Betahistine Dihydrochloride in the Treatment of Major Depression With Atypical Features
Brief Title: Pilot Study of Betahistine Dihydrochloride in the Treatment of Major Depression With Atypical Features
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Erik Nelson, Adjunct Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nelson #1
Record Dates: First submitted 2007-12-28; First posted 2008-01-03 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Recurrent Major Depressive Disorder With Atypical Features
Keywords: Depression; Betahistine Dihydrochloride
MeSH Terms: conditions — Depression | interventions — Betahistine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Betahistine dihydrochloride (Experimental): Oral betahistine dihydrochloride; daily dose 50-300 mg
  Interventions: Drug: betahistine dihydrochloride

INTERVENTIONS:
Drug: betahistine dihydrochloride — oral, 50-300 mg, daily
  Other Names: SERC

SUMMARY:
The purpose of this study is to determine a dose of the investigational drug betahistine dihydrochloride that is both well tolerated and potentially effective in treating the symptoms of atypical depression. Atypical depression is characterized by the ability of the person's mood to improve temporarily in response to positive events, as well as features such as increased appetite, increased sleep and severe fatigue.

DETAILED DESCRIPTION:
All patients will start taking 50 mg of betahistine dihydrochloride on treatment day 1 (after baseline visit). Starting on day 4, the daily dose will be increased by adding a 50 mg dose. If tolerated, the daily dose will be titrated to 200 mg. At the end of week 3, the dose will be titrated to 300 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed written informed consent
2. Be male and/or female outpatients 18 65 years of age, inclusive
3. For women: must be surgically sterile, 2 years postmenopausal, or, if they have childbearing potential, using a medically accepted method of birth control and agree to continue use of this method for at least 30 days after the last dose of study drug (i.e., barrier method with spermicide, steroidal contraceptive or intrauterine device [IUD])
4. Meet DSM IV1 criteria for major depressive episode (unipolar), with atypical features
5. Have a score of 20 or greater on the Hamilton Depression Rating, 28-item version (HAM-D-28)
6. Have a complete medical and psychiatric history, physical examination, laboratory evaluation, and ECG before study entry.
7. Have baseline laboratory values and ECG that are normal, or abnormalities that are clinically insignificant

Exclusion Criteria:

1. Have significant and/or unstable gastrointestinal, neurological, endocrine, cardiovascular, pulmonary, renal, hepatic, immunological or hematological disease; organic brain disease; or cancer as determined by history, physical, ECG, and laboratory examination
2. Have a history of peptic ulcer disease
3. Have a history of severe asthma
4. Have a current diagnosis of pheochromocytoma
5. Are pregnant, intending to become pregnant, nursing, at risk for pregnancy, or not practicing medically acceptable birth control. (A blood pregnancy test will be performed at the screening visit)
6. Meet criteria for DSM IV1 psychoactive substance abuse or dependence in the past month
7. Have a history of a psychotic disorder
8. Use any medications that, in the judgment of the investigator, might have psychotropic effects, or interact unfavorably with betahistine dihydrochloride including centrally acting antihistaminic agents
9. Have a history of hypersensitivity to betahistine dihydrochloride
10. Exhibit, or suggestion that they may display, behavior that will not be conducive to the study procedures
11. Are at significant risk of suicide as indicated by a score of 3 or greater on item number 11 on the HAM-D 28
12. Have received any investigational product within 28 days of Screening
13. Have used any antidepressant within 7 days of Screening (14 days for MAOIs; 21 days for fluoxetine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Nelson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrollment began 7/1/2007
Pre-assignment Details: 7 patients signed consent & 6 patients screen-failed
Groups:
- Betahistine Dihydrochloride: All patients start taking betahistine dihydrochloride 50 mg, which will be increased by 50 mg up to a maximum of 300 mg.
Period: Overall Study
Arm/Group | Betahistine Dihydrochloride
Started | 1
Patients Receiving Drug | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Betahistine Dihydrochloride
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerable Dose of Betahistine Dihydrochloride in mg
Description: The highest betahistine dose that is well tolerated when patients are titrated from 50 mg to a maximum 300 mg of daily divided doses.
Time Frame: 7 weeks
Population: The patient did not complete the study and not enough data were collected to be analyzed.
Arm/Group | Betahistine Dihydrochloride
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Entire Study
Arm/Group | Betahistine Dihydrochloride
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betahistine Dihydrochloride (N=1)
Mild to Moderate Gastrointestinal irritation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No